CLINICAL TRIAL: NCT06549556
Title: The Value of Using Colostrum Supplements on the Physical Performance and Cognitive Function in Healthy Subjects and Type 2 Diabetes: A Case-management Comparative Study
Brief Title: The Value of Using Colostrum Supplements on the Physical Performance and Cognitive Function in Healthy Subjects and Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Collaborators: Al-Farabi Kazakh National University (Unknown)
Responsible Party: Principal Investigator, Hayder Adnan Fawzi, Assistant Prof, Al-Rasheed University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-3672 in 27/10/2024
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Colostrum; Diabetes Mellitus, Type 2; Cognition; Physical Functional Performance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Healthy Control) (Placebo Comparator): 24 Patients receiving Placebo Capsule per oral once daily for 60 days.
  Interventions: Other: Placebo
- Group 2 (Healthy control) (Active Comparator): 26 Patients receiving Colostrum Capsule 500 mg (Colostrum® 500 mg Veg Capsules, nowfoods®, Illinois, USA), one capsule per oral once daily for 60 days.
  Interventions: Drug: Colostrum Capsule 500 mg (Colostrum® 500 mg Veg Capsules, nowfoods®, Illinois, USA)
- Group 3 (Diabetes Type 2) (Placebo Comparator): 23 Patients receiving Placebo Capsule per oral once daily for 60 days.
  Interventions: Other: Placebo
- Group 4 (Diabetes Type 2) (Active Comparator): 27 Patients Receiving Colostrum Capsule 500 mg (Colostrum® 500 mg Veg Capsules, nowfoods®, Illinois, USA), one capsule per oral once daily for 60 days.
  Interventions: Drug: Colostrum Capsule 500 mg (Colostrum® 500 mg Veg Capsules, nowfoods®, Illinois, USA)

INTERVENTIONS:
Drug: Colostrum Capsule 500 mg (Colostrum® 500 mg Veg Capsules, nowfoods®, Illinois, USA) — Brand name: (Colostrum® 500 mg Veg Capsules) capsules per oral / once daily / 60 days duration.
  Arms: Group 2 (Healthy control); Group 4 (Diabetes Type 2)
Other: Placebo — Placebo Capsule / Capsules per oral / once daily / 60 days duration
  Arms: Group 1 (Healthy Control); Group 3 (Diabetes Type 2)

SUMMARY:
The goal of this interventional Randomized clinical is to compare the effect of colostrum pharmaceutical preparation and placebo in a sample of Iraqi participants. The main questions to answer are:

1. What are the effects of the tested regimens on the level of IL-1 and IL-15.
2. What are the effects of the tested regimens on the Fasting Blood glucose?
3. What are the effects of the tested regimens on the HbA1C?
4. What are the effects of the tested regimens on the Body Mass Index?
5. What are the effects of the tested regimens on the Lipid profile?
6. What are the effects of the tested regimens on C-reactive protein?
7. What are the effects of the tested regimens on Hematological indices?
8. What are the effects of the tested regimens on Rate pressure product?

Participants will be separated into four groups:

1. Group 1 (Healthy control): 24 Patients, will be receiving Placebo Capsule per oral once daily for 60 days
2. Group 2 (Healthy control) : 26 Patients, will be receiving Colostrum Capsule 500 mg per oral once daily.
3. Group 3 (Diabetes Type 2): 23 Pateins, will be receiving Placebo Capsule per oral once daily for 60 days
4. Group 4 (Diabetes Type 2) : 27 Patients, will be receiving Colostrum Capsule 500 mg per oral once daily.

Researchers will compare Groups 1,2,3, and 4 to observe the effect of the tested treatment regimens on Fasting Blood Glucose, HbA1c, Lipid profile, Rate pressure product, C-reactive protein, Hematological indices, and Body Mass Index. and use these measures In special formulas to determine the effect of the tested regimens on physical performance and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Apperantly Healthy patients for control
* Patients diagnosed with T2DM
* Age between 18-70

Exclusion Criteria:

* Patients with T1DM
* Patients with a drug history of anabolic substances for more than 14 days duration.
* Patients with co-morbidities (e.g. CVS, renal, hepatic, and endocrine disorders)
* Pregnancy, lactation, or female patient willing for conception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Serum IL-1 Level | at Baseline, and After 60 days of treatment.
  Measured in Pg/mL
Serum IL-15 Level | at Baseline, and After 60 days of treatment.
  Measured in Pg/mL
Fasting Blood Sugar (FBS) | at Baseline, and After 60 days of treatment.
  Measured in mg/dL
Hemoglobin A1C (HbA1C) | at Baseline, and After 60 days of treatment.
  Measured in percent from total Hemoglobin
Body Mass Index (BMI) | at baseline, and after 60 days of treatment.
  Measured in Kg/m²

SECONDARY OUTCOMES:
Serum C-reactive protein (CRP) | At baseline, and after 60 days of treatment
  Measured in mg/dL
Rate Pressure Product | at Baseline, and after 60 days of treatment.
  Measured in an equation combining Heart rate in (BPM) and blood pressure in (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khalid Mohammed Albasri, MSc. Pharmacology, Principal Investigator — Al-Farabi Kazakh National University; Hayder Adnan Fawzi, PhD. Clinical Pharmacy, Study Chair — Al-Rasheed University College
Locations (1):
- Al-Zahraa Teaching Hospital, Wāsiţ, Iraq